TR Istanbul University-Cerrahpaşa ID: NYalcinbas

The Effectiveness of Motivational Interviewing in Reducing the Use of Household Chemicals and Personal Care Products During Pregnancy

**Informed Consent Form: December 30, 2023** 

Clinical Trial Number: NCT ID not yet assigned

## **INFORMED CONSENT FORM**

**Research Title**: The Effectiveness of Motivational Interviewing in Reducing the Use of Household Chemicals and Personal Care Products During Pregnancy

## Dear Participant,

You have been invited to participate in the above-mentioned research. Before agreeing to take part in this research, you should understand the purpose of the research and make your decision freely within the framework of this information. Please read the following information carefully, if you have any questions, ask and ask for a clear answer.

This research; It is carried out by graduate student Nazlı YALCINBAS under the coordination of Prof. Dr. Neslihan OZCAN, one of the faculty members of Istanbul University-Cerrahpaşa Faculty of Health Sciences, Department of Midwifery

The study will be carried out to test the effectiveness of motivational interviewing in reducing the use of household chemicals and personal care products during pregnancy. The motivational interview method is an interview method used to give people healthy behaviors. In accordance with the criteria for inclusion in the study, some of the participants will be assigned to the experimental group and some to the control group. You will be informed by the researcher which group you are assigned to. Motivational interviews will be held with all participants selected for the experimental group to reduce the use of household chemicals and personal care products. In this context, face-to-face meetings will be held 2 times in total, lasting an average of 30-45 minutes, by determining the time interval in which the researcher and the participant are suitable. One month after the interviews, the form applied at the beginning of the research will be applied again. Participants in the control group will be given an informative brochure. If they wish, the same interviews can be carried out with the participants who make up the control group after the end of the research.

Your participation in the research is entirely voluntary and you have the right to refuse to participate in the research. You can leave the research at any time. You will not incur any financial liability by participating in this research. In addition, you will not be paid anything. If you withdraw from the research or are removed from the research by the researcher, the data about you will not be used. However, once the data is anonymized, you will not be able to withdraw from the research. All information obtained from you will be kept confidential, and the confidentiality of your credentials, if any, will be maintained when the research is published.

"I read (or listened orally) to the text above, which contains information that should be given to volunteers before starting the research. I asked my questions to the researchers on the issues that I thought were missing and received satisfactory answers. I believe that I have fully understood all the explanations presented to me in written and oral form. I was given enough time to decide whether I wanted to participate in the study. Under these circumstances, I declare that I accept the use of personal information obtained within the scope of the research for scientific purposes, its presentation and dissemination provided that the rules of confidentiality are complied with, without any pressure or coercion, of my own free will."

| | | | History | Signature |
|-------------------------------|------|-----|---------|-----------|
| Participant name and surname: | | | | |
| Researcher's | name | and | | |

| surname: |
|--------------------|
| Interview witness: |